CLINICAL TRIAL: NCT03403478
Title: Effects of Aquatic Exercise on Post-exercise Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Collaborators: University Center of Joao Pessoa - UNIPE (Unknown)
Responsible Party: Principal Investigator, Bruno Teixeira Barbosa, Assistant Professor, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 79609117.0.0000.5188
Record Dates: First submitted 2018-01-07; First posted 2018-01-18 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Hypertension; Aging; Obesity
Keywords: Hemodynamics; Aquatic exercise; Elderly
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: To acute session, the participant will not be informed about what aquatic exercise session (light-, moderate-, high-intensity or control) intensity will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (No Intervention): The volunteers will be instructed to remain in an orthostatic position immersed in water up to the imaginary line of the xiphoid process for 45 minutes without performing jerky body movements.
- LICE (Experimental): The light-intensity continuou exercise (LICE) session comprises a 45-minute of guide walking into the pool at 55-60% of maximum heart rate (HRmax). The HR will be checked every 2 minutes during the whole session.
  Interventions: Other: LICE
- MICE (Experimental): The moderate-intensity continuous exercise (MICE) will bem performed divided into 3 phases: warm-up (10 minutes), main part (30 minutes) and cool down (5 minutes). The warm-up and cool down will be performed at 55-60% HRmax. The main part will last 30 minutes and will be performed by 3 sets of 5 exercises lasting 2 minutes each one at 70-75% HRmax. For all phases, HR will be measured every 2 minutes during the whole session.
  Interventions: Other: MICE
- HIIE (Experimental): The high-intensity intervaled exercise (HIIE) will bem performed divided into 3 phases: warm-up (10 minutes), main part (15 minutes) and cool down (5 minutes). The warm-up and cool down will be performed at 55-60% HRmax. The main part will last 15 minutes and will be performed by 2 sets of 5 exercises lasting 30 seconds to each exercise combined with 1 minute of active recovery. The exercise moment will be performed at 80-85% HRmax and the 1-minute active recovery at 55-60% HRmax. For both warm-up and cool down, HR will be measured every 2 minutes. For main part, HR will be measured at the end of each 30-seconds from exercise.
  Interventions: Other: HIIE
- Aquatic exercise training (Experimental): The participants will be submitted to a 12-weeks of aquatic exercise program, twice a week, for 1 hour each day.
  Interventions: Other: Aquatic exercise training

INTERVENTIONS:
Other: LICE — No specific exercise will be performed. The participant will walk into the pool accompanied with a researcher for 45 minutes.
  Arms: LICE
Other: MICE — The following exercises will be carried out: a) jumping jacks (shoulder abduction and adduction); b) horizontal adduction and abduction of the shoulder; c) stationary running with knee elevation; d) pull and push horizontally with upper limbs; e) pull and push vertically with upper limbs.
  Note: For exercises 'a' and 'b', the legs alternated in movements in the sagittal plane to provide greater stability to the participant's movement. For exercises 'd' and 'e', the legs simulates a stationary running.
  Arms: MICE
Other: HIIE — The following exercises will be carried out: a) jumping jacks (shoulder abduction and adduction); b) horizontal adduction and abduction of the shoulder; c) stationary running with knee elevation; d) pull and push horizontally with upper limbs; e) pull and push vertically with upper limbs.
  Note: For exercises 'a' and 'b', the legs alternated in movements in the sagittal plane to provide greater stability to the participant's movement. For exercises 'd' and 'e', the legs simulates a stationary running.
  Arms: HIIE
Other: Aquatic exercise training — The sessions of the aquatic exercise training will be divided into 3 phases: warm-up (10 minutes), main part (40 minutes) and cool down.
  In order to increase intensity to aquatic exercise, the training program will carried out as follows:
  From week 1 to 4 the instructors will use a 128 bpm musics in both warm-up and cool down. In main part, will be used a 130 bmp musics.
  From week 5 to 8 the instructors will use a 130 bpm musics in both warm-up and cool down. In main part, will be used a 132 bmp musics.
  From week 9 to 12 the instructors will use a 132 bpm musics in both warm-up and cool down. In main part, will be used a 135 bmp musics.
  Arms: Aquatic exercise training

SUMMARY:
This is a randomized controlled trial. The present study involves an acute and chronic intervention, which is a water-based exercise (one session: to acute intervention; 12-weeks of aquatic exercise program: to chronic intervention). The sample will be composed by elderly enrolled in university extension program titled "Hidroginastica na Terceira Idade" (Hydrogymnastics in aging). It will be evaluated the effects of water-based exercise on hemodynamics, self-reported sleep quality, depressive symptoms, quality of life, body composition, level of physical activity and functional capacity. The investigators hypothesized that an acute water-based exercise under different intensities promotes hemodynamics changes in elderly. In addition, the investigators hypothesized that 12-weeks of aquatic exercise may lead improvements in self-reported sleep quality, depressive symptoms, quality of life, body composition, level of physical activity and functional capacity in elderly.

ELIGIBILITY:
Inclusion Criteria:

* Elderly (60 years and over)
* Able to practice physical exercise in water
* Able to answer all questionnaires
* Non-smoker

Exclusion Criteria:

* Morbid obese
* Those who not complete all data collection procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Entire day (an average of 24 hours).
  The blood pressure will be measured by a Ambulatory Blood Pressure Monitoring (ABPM).
Blood pressure | Up to 1 hour post-exercise session
  The blood pressure will be measured by an automatic blood pressure device (OMRON HEM-720).

SECONDARY OUTCOMES:
Self-reported sleep quality | Approximately 15 minutes
  Pittsburgh Sleep Quality Index
Depressive symptoms (Mental disorders) | Approximately 5 minutes
  Geriatric depressive symptoms (GDS-15) is a validated questionnaire which will be used in order to evaluate depressive symptoms in elderly.
Self-reported quality of life | Approximately 15 minutes
  Quality of life will be assessed by the WHOQOL-OLD questionnaire and it consists of 24 items on the likert scale attributed to 6 facets: 1) Sensory functioning, 2) Autonomy, 3) Past, present and future activities, 4) Social participation, 5) Death and dying, and 6) Intimacy. Each facet is composed of 4 items, so for each facet the score can range from 4 to 20. For this evaluation, the higher the score, the higher the quality of life.
Level of physical activity (BAECKE modified to elderly) | Approximately 5 minutes
  The Habitual Physical Activity Questionnaire originated in 1982 by Baecke and colleagues (BAECKE; BUREMA, FRIJTERS, 1982) and was adapted for the elderly and validated later (VORORRIPS et al., 1991) and recently translated into Portuguese (SIMÕES, 2009). It is applied in the form of an interview, and has as reference the last 12 months being divided into 3 sections (1 - Domestic physical activities, 2 - Sporting activities and 3 - Activities in free time). From the scores attributed to each response provided by the elderly, scores equivalent to each section cited above are established. It is suggested that 3 cutoff points be created for the classification of the elderly regarding the level of physical activity (low, moderate and high) based on terciles.
Functional Capacity | Approximately 35 minutes
  AAPHERD test battery

CONTACTS AND LOCATIONS:
Overall Officials: Bruno T Barbosa, Master, Principal Investigator — University Center of Joao Pessoa - UNIPE
Locations (1):
- Bruno Teixeira Barbosa, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No